CLINICAL TRIAL: NCT00177983
Title: Support to Patients and Families
Brief Title: Web-based Support for People With Schizophrenia and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: R01MH063484 (NIH); R01MH063484 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Relapse Rates Related to Website Usage
Keywords: Schizophrenia; Relapse; Psychological distress
MeSH Terms: conditions — Schizophrenia; Recurrence

INTERVENTIONS:
Behavioral: (relapse rate)

SUMMARY:
This study will assess the feasibility of using the internet and in-home computers to provide advice from health care professionals, social support, and health information to people with schizophrenia and their families.

DETAILED DESCRIPTION:
The objective of this study is to assess the feasibility of using the World Wide Web (Web) and in-home computers to provide patients suffering from schizophrenia and their families advice from health care professionals, social support, and information.

The purposes of this intervention are to improve: 1) the availability, convenience and use of needed mental health services; 2) family support for their ill family members; and 3) patient and family outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia Able to speak and read English Regular contact with a family member

Exclusion Criteria:

* Enrolled in another study

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80
Dates: Start 2003-01; Study Completion 2005-01

PRIMARY OUTCOMES:
The outcome, patient relapse, will be assessed for the patients in the intervention group and control group by estimating the size of the intervention's effect on relapse rate.

SECONDARY OUTCOMES:
For the primary caregiver, the distribution of the psychological distress measure will be examined and transformation will be made if necessary for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Armando J Rotondi, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States